CLINICAL TRIAL: NCT03739762
Title: Randomized Trial to Reduce Sitting Time and Improve Cardiometabolic Health in Obese Older Adults
Brief Title: Healthy Aging Resources to Thrive (HART)
Acronym: HART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1315055-1; 1R01HL132880-01A1 (NIH)
Record Dates: First submitted 2018-10-31; First posted 2018-11-14 (Actual); Results first posted 2023-12-05 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-05

CONDITIONS: Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of two cohorts/arms: one called "i-STAND" with coaching sessions focused directly on sitting less and standing more; the other called "Healthy Living" with coaching sessions focused on various topics related to a healthy lifestyle, but without a focus on standing more. Those randomized to the i-STAND intervention will also be re-randomized half-way through the study, with half of that cohort moving on to phase 2, which involves booster sessions on sitting less and standing more. All participants regardless of cohort will be mailed a blood pressure monitor and a scale to keep. UPDATE: As of March 31, 2022, beginning in our final year (year 5) of the study, participants randomized to the i-STAND intervention will no longer be re-randomized at 6 months. We will no longer follow participants to the 12-month timepoint and will end all activities after the 6-month timepoint.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- i-STAND (Experimental): i-STAND participants have a Baseline visit followed by the 1st Coaching visit. They receive wristbands that vibrate every 15 minutes to prompt a standing break, standing desks, workbook & 10 phone-based coaching calls focused on sitting less/standing more. There is a 3 month measurement visit. Program ends at 6 months when they wear an activPAL & have a measurement visit. Coach provides feedback on activPAL sitting time after all activPAL wears (Bsln, 3, 6 & 12 month). They may opt to wear activPAL at 6 weeks & get feedback. They are re-randomized at 6 months; half to be assigned to intervention boosters (5 more phone sessions/a 9-month optional activPAL) before the 12 month final activPAL & final measurement visit. Those not randomized to boosters will have no contact until the 12 month visit. UPDATE: As of 3/31/2022, (final year 5), i-STAND ppts will no longer be re-randomized at 6 months. We will no longer follow to the 12-month timepoint & will end all activities after 6-months.
  Interventions: Behavioral: i-STAND
- Healthy Living control (Active Comparator): In this arm, participants have a phone-based Baseline visit followed by the 1st phone-based Coaching visit. No prompting devices/desks are offered; coaching focuses on topics related to healthy living, but with no focus on sitting less/standing more. They have 10 phone calls with a health coach. Participants receive a workbook. All content is from KaiserPermanente WA and is available to all members. Participants select topics & review them with their health coach. At 3 months, participants have a measurement visit. The program ends at 6 months where participants will wear an activPAL and have a measurement visit. After that, there is no contact with the study team until 12 months when they will again wear an activPAL & have a final measurement visit. UPDATE: As of 3/31/2022, our final year (year 5) of the study, participants randomized to the control arm will no longer be followed to the 12-month timepoint and will end all activities after the 6-month timepoint.
  Interventions: Other: Healthy Living control

INTERVENTIONS:
Behavioral: i-STAND — Via in-person and phone coaching sessions, participants randomized to this arm will be coached to find ways to sit less and stand more, and look for ways to change their home environment to encourage this, as well as look at how their lifestyle may contribute to their sitting time. Participants in this arm may be re-randomized at the half-way point to continue with additional phone coaching sessions. (As of 3/31/2022 Re-randomizations are no longer taking place)
  Arms: i-STAND
Other: Healthy Living control — In this arm, participants will have phone coaching sessions focused on a variety of topics aimed at improving healthy habits. There is no focus on standing more or sitting less.
  Arms: Healthy Living control

SUMMARY:
Healthy Aging Resources to Thrive (HART) uses a rigorous two-stage randomized control design, adapted and refined based on pilot studies, to test a novel intervention to reduce sitting time in older adults. Half the participants will be randomized to the intervention aimed at decreasing sitting time, and the other half will be randomized to a healthy living control that does not focus on reduced sitting time. After 6 months, the intervention group will be further randomized so that half continue with the intervention and the other half receive no further intervention. All participants will be followed for 12 months.

DETAILED DESCRIPTION:
Healthy Aging Resources to Thrive (HART) is a two-stage randomized controlled trial (RCT) of adults over age 60 with obesity to determine the efficacy of a novel sitting-reduction intervention and its impact on cardiometabolic risk markers. Participants will be randomized to a 6-month sitting reduction intervention (termed I-STAND) or healthy-living attention control (Stage 1). All participants will be mailed a scale and a blood pressure monitor (to keep) which will be used during the phone-based measurement visits at Baseline, 3, 6 and 12 months. All participants will have phone-based Coaching sessions.

After 6 months, I-STAND participants will be re-randomized to receive either booster sessions or no further intervention (Stage 2). Attention control participants will receive no further intervention. All participants will be followed for 12 months total with phone-based assessments at baseline, 3, 6, and 12 months. Primary outcomes are reduction in sitting time at 6 months, objectively measured using the activPAL device, and blood pressure. The design will answer novel questions about the impact of sitting reduction on cardiometabolic risk markers as well as maintenance of sitting reduction.

UPDATE: As of 3/31/31, (final year 5) of the study, participants randomized to the i-STAND intervention will no longer be re-randomized at 6 months. We will no longer follow participants to the 12-month timepoint & will end all activities after 6-months.

ELIGIBILITY:
Inclusion Criteria: • Self-reported sitting time of 6+ hours per day

* BMI ≥30 and <50 kg/m2
* men and women of all races and ethnicities from anywhere in the KPWA region (state-wide)
* We will oversample people of color statewide
* Able to walk one block
* Able to speak and read English,
* no self-reported vision limitations, sedentary time, use of an assistive device, able to stand.
* no cognitive impairment that is perceived by the study staff during phone screening
* Willingness to wear device (activPAL)
* Willingness to participate in study for a full year
* Continuously enrolled at KP for previous 12 months
* Not on the No Contact list
* Not previously enrolled in ISTAND or TABS
* Not currently enrolled in ACT, STOP-FALLS or SMARRT studies

Exclusion Criteria:

* unable to speak and read English (phone screen)
* unable to walk 1 block (with or without assistive devices) (phone screen)
* self-reported sitting time less than 6 hours per day (phone screen)
* diagnosis codes indicating hearing loss, dementia or serious mental illness (e.g., schizophrenia, bipolar disorder), or a terminal or serious illness (e.g., cancer) in the past 2 years (from the EMR)

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dori E Rosenberg, PhD, MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Rosenberg DE, Greenwood-Hickman MA, Zhou J, Cook AJ, Mettert KD, Cooper J, Arterburn D, Green BB, Walsh-Bailey C, Kerr J, Owen N, Dunstan D, McClure JB. Protocol for a randomized controlled trial of sitting reduction to improve cardiometabolic health in older adults. Contemp Clin Trials. 2021 Dec;111:106593. doi: 10.1016/j.cct.2021.106593. Epub 2021 Oct 16. PMID 34666182
- [Background] Greenwood-Hickman MA, Dahlquist J, Cooper J, Holden E, McClure JB, Mettert KD, Perry SR, Rosenberg DE. "They're Going to Zoom It": A Qualitative Investigation of Impacts and Coping Strategies During the COVID-19 Pandemic Among Older Adults. Front Public Health. 2021 May 19;9:679976. doi: 10.3389/fpubh.2021.679976. eCollection 2021. PMID 34095079
- [Result] Greenwood-Hickman MA, Zhou J, Cook A, Mettert KD, Green B, McClure J, Arterburn D, Florez-Acevedo S, Rosenberg DE. Exploring Differences in Older Adult Accelerometer-Measured Sedentary Behavior and Resting Blood Pressure Before and During the COVID-19 Pandemic. Gerontol Geriatr Med. 2022 Apr 27;8:23337214221096007. doi: 10.1177/23337214221096007. eCollection 2022 Jan-Dec. PMID 35506125
- [Result] Rosenberg DE, Zhu W, Greenwood-Hickman MA, Cook AJ, Florez Acevedo S, McClure JB, Arterburn DE, Cooper J, Owen N, Dunstan D, Perry SR, Yarborough L, Mettert KD, Green BB. Sitting Time Reduction and Blood Pressure in Older Adults: A Randomized Clinical Trial. JAMA Netw Open. 2024 Mar 4;7(3):e243234. doi: 10.1001/jamanetworkopen.2024.3234. PMID 38536177
- [Derived] Florez-Acevedo S, Greenwood-Hickman MA, Zhu W, Cook AJ, Delaney K, Green BB, Arterburn DE, McClure JB, Rosenberg DE. Exploratory Analysis of Mental Health and Quality of Life Outcomes in a Randomized Controlled Trial to Reduce Sitting Time in Older Adults With Obesity. J Aging Phys Act. 2025 Nov 12:1-12. doi: 10.1123/japa.2024-0387. Online ahead of print. PMID 41223847

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Goal was 284 randomized participants. A total of 357 potential participants were recruited, with 283 consenting and completing baseline measurements and randomization.
Pre-assignment Details: We had 11 participants consent* to the study but who were never randomized thus *not enrolled*. Of these, 3 completed a baseline visit but before randomization, 2 never responded to our attempts to reach them (5 calls and one letter) and 1 said they were too busy to continue. The remaining 8 were non responsive to our attempts to reach them after initial consent.
  All of these participants were remote and thus their randomization took place up to 2 weeks after the baseline visit.
Period: Overall Study
Arm/Group | i-STAND | Healthy Living Control
Started | 140 | 143
Completed | 137 | 136
Not Completed | 3 | 7
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | i-STAND | Healthy Living Control | Total
Number analyzed (Participants) | 140 | 143 | 283
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 46 | 89
  >=65 years | 97 | 97 | 194
Age, Continuous [Mean (Full Range); unit: years] | 68.57 [60 to 88] | 69.03 [60 to 86] | 68.8 [60 to 88]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Non-Binary | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 99 | 187
  Male | 52 | 44 | 96
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 4 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 4 | 2 | 6
  Black or African American | 25 | 17 | 42
  White | 97 | 107 | 204
  More than one race | 7 | 7 | 14
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants] — Pre-pandemic participants were recruited from King County, WA. With the onset of the pandemic and the switch to a 100% remote study, we expanded statewide.
  Participants
    United States | 140 | 143 | 283
Baseline Measure of Time Spent Sitting or Lying Down [Mean (Standard Deviation); unit: Minutes] — Baseline sitting time in minutes was measured using the activPAL device (does not include sleep time). Population: We had missing data for baseline sitting time: 2 in the intervention group and 4 in the control group.
  Minutes
    number analyzed (Participants) | 138 | 139 | 277
    (all) | 650.4 (117.9) | 654.5 (115.5) | 652.4 (116.5)
Baseline Measure of Systolic Blood Pressure mmHg [Mean (Standard Deviation); unit: mmHg] — Population: We had missing SBP for 1 participant in the baseline control group
  mmHg
    number analyzed (Participants) | 140 | 142 | 282
    (all) | 135.4 (18.8) | 136.7 (18.3) | 136.1 (18.5)
Baseline measure of Diastolic Blood Pressure mmHg [Mean (Standard Deviation); unit: mmHg] — Population: We had missing DBP for 1 participant in the baseline control group
  mmHg
    number analyzed (Participants) | 140 | 142 | 282
    (all) | 79.6 (11.1) | 79.8 (10.2) | 79.7 (10.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Time Spent Sitting or Lying Down at 6 Months
Description: Time (minutes) spent sitting/lying during waking hours will be measured objectively by the activPAL worn for one week following each measurement visit.
Time Frame: Change from Baseline at 6 months
Population: Number of participants who had a 6-month measure for change in sitting time
Measure: Mean (95% Confidence Interval); unit: Minutes
Arm/Group | i-STAND | Healthy Living Control
Number analyzed (Participants) | 124 | 122
Minutes | -40.36 [-54.86 to -25.85] | -8.51 [-23.97 to 6.95]
Statistical Analysis 1: Comparison: i-STAND vs Healthy Living Control; The sample size of 284 ensured 90% power to detect a 41-minute difference in sitting time between I-STAND and the attention control from baseline to 6 months, assuming a standard deviation (SD) of 97 minutes/day for change in sitting time (based on our pilot data), and 15% loss to follow-up. Sample and power calculations were performed using R software version 3.5 [39] via simulation, assuming specified SDs and differences between means; Test type: Superiority; p = 0.003, Regression, Linear; The model fit was a linear regression model with GEE on the outcome change from baseline; Mean Difference (Final Values) = -31.85, 95% CI 2-sided [-52.91 to -10.79]

2. Primary Outcome: Change in SystolicBlood Pressure at 6 Months
Description: Another primary outcome is change in systolic blood pressure. This will be measured at the measurement visits using blood pressure monitors mailed to the participant
Time Frame: Change from Baseline at 6 months
Population: Number of participants who had a 6-month measure for SBP
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | i-STAND | Healthy Living Control
Number analyzed (Participants) | 127 | 127
mmHg | -6.67 [-8.82 to -4.52] | -3.19 [-5.44 to -0.94]
Statistical Analysis 1: Comparison: i-STAND vs Healthy Living Control; Test type: Superiority; p = .033, Regression, Linear; The model fit was a linear regression model with GEE on the outcome change from baseline; Mean Difference (Final Values) = -3.48, 95% CI 2-sided [-6.68 to -0.28]

3. Primary Outcome: Change in Diastolic Blood Pressure at 6 Months
Description: Another primary outcome is change in diastolic blood pressure
Time Frame: Change from Baseline at 6 months
Population: Number of participants who had a 6-month measure for Diastolic BP
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | i-STAND | Healthy Living Control
Number analyzed (Participants) | 127 | 127
mmHg | -1.32 [-2.66 to 0.02] | -1.58 [-2.93 to -0.23]
Statistical Analysis 1: Comparison: i-STAND vs Healthy Living Control; Test type: Superiority; p = .784, Regression, Linear; The model fit was a linear regression model with GEE on the outcome change from baseline; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-1.63 to 2.16]

4. Secondary Outcome: Change in Weight at 6 Months
Description: Participants provide their weight at each measurement visit. Weight is measured in pounds using a scale mailed to the participant.
Time Frame: Change from Baseline at 6 months
Measure: Mean (95% Confidence Interval); unit: pounds
Arm/Group | i-STAND | Healthy Living Control
Number analyzed (Participants) | 99 | 111
pounds | -3.56 [-5.50 to -1.63] | -3.45 [-4.95 to -1.94]
Statistical Analysis 1: Comparison: i-STAND vs Healthy Living Control; Test type: Superiority; p = .927, Regression, Linear; The model fit was a linear regression model with GEE on the outcome change from baseline; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-2.61 to 2.38]

5. Secondary Outcome: Change in BMI at 6 Months
Description: BMI was calculated as [weight in kg]/[height in m]2.
Time Frame: Change from Baseline at 6 months
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | i-STAND | Healthy Living Control
Number analyzed (Participants) | 99 | 111
kg/m^2 | -0.51 [-0.85 to -0.17] | -0.54 [-0.81 to -0.26]
Statistical Analysis 1: Comparison: i-STAND vs Healthy Living Control; Test type: Superiority; p = .916, Regression, Linear; The model fit was a linear regression model with GEE on the outcome change from baseline; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.42 to 0.47]

6. Secondary Outcome: Change in Waist Circumference at 6 Months
Description: Participants provided their waist circumference at each measurement visit. Waist circumference was measured at the superior border of the iliac crest.
Time Frame: Change from Baseline at 6 months
Measure: Mean (95% Confidence Interval); unit: inches
Arm/Group | i-STAND | Healthy Living Control
Number analyzed (Participants) | 124 | 124
inches | -1.0 [-1.55 to -0.45] | -0.64 [-1.09 to -0.19]
Statistical Analysis 1: Comparison: i-STAND vs Healthy Living Control; Test type: Superiority; p = .325, Regression, Linear; The model fit was a linear regression model with GEE on the outcome change from baseline; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-1.09 to 0.36]

ADVERSE EVENTS:
Time Frame: 6 months
Description: AE data was collected at coaching calls and measurement calls no matter the relation to the study. Adverse Events were monitored/assessed without regard to the specific Adverse Event Term.
Arm/Group | i-STAND | Healthy Living Control
All-Cause Mortality (participants affected / at risk) | 0/140 | 0/143
Serious Adverse Events (participants affected / at risk) | 6/140 | 6/143
Other Adverse Events (participants affected / at risk) | 72/140 | 47/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | i-STAND (N=140) | Healthy Living Control (N=143)
Unrelated SAE (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — Unrelated to study
Unrelated SAE (Cardiac disorders) | 0 (0) | 1 (1) — Unrelated to study
Unrelated SAE (Eye disorders) | 1 (1) | 0 (0) — Unrelated to Study
Unrelated SAE (Gastrointestinal disorders) | 1 (1) | 0 (0) — Unrelated to Study
Unrelated SAE (General disorders) | 0 (0) | 1 (1) — Unrelated to Study
Unrelated SAE (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — Unrelated to Study
Unrelated SAE (Renal and urinary disorders) | 2 (2) | 0 (0) — Unrelated to Study
Unrelated SAE (Surgical and medical procedures) | 0 (0) | 1 (1) — Unrelated to Study
Unrelated SAE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Unrelated to Study
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | i-STAND (N=140) | Healthy Living Control (N=143)
Unrelated Other AE (General disorders) | 14 (14) | 12 (12)
Unrelated Other AE (Musculoskeletal and connective tissue disorders) | 35 (35) | 19 (19)
Anticipated Related AE (Skin and subcutaneous tissue disorders) | 9 (9) | 1 (1) — These are expected and related to wearing the device adhered to the skin with Tegaderm (potential skin irritant)
Unrelated Other AE (Vascular disorders) | 14 (14) | 15 (15)

LIMITATIONS AND CAVEATS:
Limitations of our study include the interruption caused by the COVID-19 pandemic, which occurred after 100 of the 283 participants were enrolled. We had to rely on participant-measured outcomes post-pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT03739762/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/62/NCT03739762/ICF_001.pdf